CLINICAL TRIAL: NCT04766047
Title: The Effect of Dexmedetomidine on the Incidence of Acute Kidney Injury in EVAR
Brief Title: The Effect of Dexmedetomidine on Kidney Function in EVAR
Acronym: DEVAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of anesthesiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Dexmedetomidine in EVAR
Record Dates: First submitted 2021-02-02; First posted 2021-02-23 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Acute Kidney Injury; Dexmedetomidine; Endovascular Aortic Repair
Keywords: Acute kidney injury, Dexmedetomidine, EVAR
MeSH Terms: conditions — Acute Kidney Injury | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEXMEDETOMIDINE AND AKI (Active Comparator): The patients of the group undergoing EVAR under general anesthesia will receive dexmedetomidine intraoperatively.
  Interventions: Drug: Dexmedetomidine
- CONTROL AND AKI (No Intervention): The patients of the group undergoing EVAR under general anesthesia will not receive dexmedetomidine intraoperatively.

INTERVENTIONS:
Drug: Dexmedetomidine — Administration of dexmedetomidine intraoperatively
  Arms: DEXMEDETOMIDINE AND AKI

SUMMARY:
This study will investigate the effect of dexmedetomidine on the incidence of postoperative acute kidney injury in patients undergoing EVAR under general anesthesia

DETAILED DESCRIPTION:
This study will compare the incidence of AKI after elective EVAR conducted under general anesthesia with and without administration of dexmedetomidine. The AKI will be evaluated through measuring NGAL and c-cystatin.

ELIGIBILITY:
Inclusion Criteria:

* elective EVAR under general anesthesia
* adult patients 18- 85 years old
* American society of anesthesiologists (ASA) physical status I - IV

Exclusion Criteria:

* refusal to participate or sign the informed consent form
* GFR < 50ml/mim
* Bradyarrhythmia <50/min
* Hemodynamic instability
* Known allergy to Dexmedetomidine
* Severe hepatic insufficiency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Kidney Injury | 1st Postoperative Day
  Assess the incidence of Acute Kidney Injury after the administration of dexmedetomine

SECONDARY OUTCOMES:
Incidence of postoperative ICU admission | Operation day to 5th postoperative day
  Record the incidence of unanticipated postoperative ICU admission
Incidence of arrhythmia | Up to 24 hours after surgery
  Record the incidence of arrhythmia postoperatively
Incidence of Postoperative Delirium | Operation day to 4th postoperative day
  Record the incidence of Postoperative Delirium postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, MD, PhD, Study Chair — University of Thessaly; Konstantinos Stamoulis, MD, PhD, Principal Investigator — University Hospital of Larissa
Locations (1):
- Univeristy of Thessaly, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No